CLINICAL TRIAL: NCT03849417
Title: PET-MRI Biomarkers of Pathological Brain Aging in Late-life Depression
Brief Title: Brain Imaging Biomarkers of Pathological Brain Aging in Late-life Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S61968
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2023-11

CONDITIONS: Depression
Keywords: Late-life depression; Electroconvulsive therapy; Neuroimaging; Aging
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood

GROUPS / COHORTS (3):
- Late-life Depression: Patients aged over 60 years old with severe depression
- Late-life Depression (ECT): Patients aged over 60 years old with severe depression who are referred for treatment with electroconvulsive therapy
  Interventions: Other: ECT
- Healthy Controls: Healthy volunteers over 60 years old who will form a comparison group

INTERVENTIONS:
Other: ECT — ECT administered as part of normal clinical management
  Groups: Late-life Depression (ECT)

SUMMARY:
This study investigates the relationships and differences in PET-MRI brain imaging biomarkers of abnormal aging and behavioral measures in late life depression compared to healthy controls, and evaluates relationships and differences in the same imaging and behavioral measures following electroconvulsive therapy. The study tests the hypotheses that late-life depression will be associated with higher levels of accelerated aging and brain disease biomarkers, and that electroconvulsive therapy works by stimulating the reorganization of brain tissue.The data collected with contribute to improved knowledge about the neurobiology of late-life psychopathology and its treatment.

DETAILED DESCRIPTION:
This clinical study is a combined single-center, cohort study with a (1) cross-sectional arm evaluating relationships and differences in PET-MR imaging and behavioral measures in 64 patients with late life depression (LLD) compared to 64 healthy controls, and (2) a longitudinal arm evaluating relationships and differences in imaging and behavioral measures in 20 patients receiving ECT as part of their normal clinical management. The study will utilise three PET tracers: (1) [11C]UCB-J, which targets the Synaptic Vesicle Glycoprotein 2A receptor, to estimate synaptic density (2) [18F]MK-6240, which targets tau associated with neurofibrillary tangles, to assess the presence of tau pathology and (3) [18F]-Flutemetamol, which targets beta-amyloid neuritic plaques in the brain, to assess the presence of cerebral amyloidosis. The main aim of the study is to clarify how hippocampal synaptic density, tau, amyloid and white matter lesions, relate to neuropsychological function, stress and ECT in late life depression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of late-life depression according to DSM 5 (patients only)
* Age over 60 years old
* Judged to be in good physical health by the investigator on the basis of medical history

Exclusion Criteria:

* history or evidence of psychiatric disease, as assessed by clinical interview (healthy controls only).
* history of major other neurological disorder, or major internal pathology that may make him/her unfit for participation according to the interpretation by the investigator (including cardiac, lung, haematological, gastro-intestinal disorders or cancer);
* current user (including ''recreational use'') of any illicit drugs,including cannabis, or has a history of drug or alcohol abuse;
* had exposure to ionizing radiation (> 1 mSv) in other research studies within the last 12 months;
* has a contra-indication for MRI scanning;
* suffers from claustrophobia or cannot tolerate confinement during PET-MRI scanning procedures; cannot lie still for 60 minutes inside the scanner;
* does not understand the study procedures
* unwilling or unable to perform all of the study procedures, or is considered unsuitable in any way by the principal investigator;
* underwent ECT within the last 3 months before enrollment (patients)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A consecutive series of hospital in-patients with late-life depression will be recruited from the Department of Old Age Psychiatry within the University Psychiatric Center, KU Leuven, Belgium. Healthy controls will be recruited from the community by researchers affiliated with the Department of Old Age Psychiatry Department & Translational Neuropsychiatry using traditional means e.g. flyer. All participants will provide written informed consent prior to enrollment in the study in accordance with the Declaration of Helsinki.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Relationship between synaptic density and hippocampal volume in LLD | 1 day
  Cross-sectional association between [11C]UCB-J binding (SUVR) and MRI-based assessment of hippocampal volume
Relationship between tau and hippocampal volume in LLD | 1 day
  Cross-sectional association between [18F]MK-6240 binding (SUVR) and MRI-based assessment of hippocampal volume
Relationship between tau and white matter (wm) pathology in LLD | 1 day
  Cross-sectional association between [18F]MK-6240 binding (SUVR) and MRI measures of white matter pathology (T2-FLAIR WMH/lesions, diffusion MRI measures in temporal lobe tracts)
Effect of tau on medial temporal neural responses to emotional stimuli and functional connectivity in LLD | 1 day
  Cross-sectional association between [18F]MK-6240 binding (SUVR), fMRI based assessment of the emotion positivity effect, and fMRI derived resting state brain networks.
Relationship between medial temporal pathology and stress | 1 week
  Association between [18F]MK-6240 binding (SUVR), hippocampal volume (MRI) and reactivity to stress (EMA) and wristband monitoring of heart rate and skin conductance.
Relationship between hippocampal volume increase following ECT and changes in synaptic density and tau | 8 weeks
  Association between change in [11C]UCB-J and [18F]MK-6240 binding (SUVR) and MRI-based assessment of hippocampal volume one week following last ECT
Amyloid changes following ECT | 8 weeks
  Change in [18F] Flutemetamol one week following the last ECT treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Vandenbulcke, MD, PhD, Principal Investigator — UZ Leuven / UPC-KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
The nature of anonymized IPD data that may be made available will be determined on an ad hoc basis and in adherence with the terms of the informed consent provided by the participants and advice from the local ethics committees and university technology transfer office.

REFERENCES:
- [Derived] Van Cauwenberge MGA, Vande Casteele T, Laroy M, Vansteelandt K, Van den Stock J, Bouckaert F, Emsell L, Vandenbulcke M. Motor dysfunction in late life depression: A mood or movement disorder? J Affect Disord. 2025 Jul 15;381:680-691. doi: 10.1016/j.jad.2025.04.053. Epub 2025 Apr 9. PMID 40203967
- [Derived] Emsell L, Laroy M, Van Cauwenberge M, Vande Casteele T, Vansteelandt K, Van Laere K, Sunaert S, Van den Stock J, Bouckaert F, Vandenbulcke M. The Leuven late life depression (L3D) study: PET-MRI biomarkers of pathological brain ageing in late-life depression: study protocol. BMC Psychiatry. 2021 Jan 28;21(1):64. doi: 10.1186/s12888-021-03063-y. PMID 33509135